CLINICAL TRIAL: NCT01056731
Title: A 16-week, Prospective, Open Label, Multicenter Study to Evaluate the Effectiveness and Safety of Rasilez® (Aliskiren) Monotherapy or in Addition With Hydrochlorothiazide 12.5 mg or 25 mg in Patients With Hypertension Stage I and II
Brief Title: A Clinical Study With Aliskiren Alone or in Combination Therapy With Diuretic Hctz in Venezuelan Hypertensive Patients.
Acronym: ANDROMEDA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPP100AVE01
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: High Blood Pressure
Keywords: high blood pressure; aliskiren; hydrochlorothiazide; control rate
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aliskiren and Aliskiren_HCTZ (Experimental): aliskiren 150 mg and 300 mg Hydrochlorothiazide 12.5 mg 25 mg
  Interventions: Drug: Aliskiren and HCTZ

INTERVENTIONS:
Drug: Aliskiren and HCTZ — Aliskiren 150 mg and 300 mg Hydrochlorothiazide 12.5 mg and 25 mg

SUMMARY:
This is an open-label, not controlled, sequential, dose escalation study of 16 weeks' duration. The study is composed of two periods: a 0-2 week optional wash-out period depending on previous antihypertensive treatment(s), followed by a 16-week open-label active treatment period. Patients will be evaluated every 4 weeks during period 2. Treatment will start with Aliskiren 150 mg with dose titration to Aliskiren 300 mg, and addition of HCTZ 12,5 mg and 25 if control of BP is not achieved (< 140/90 mmHg or 130/ 80 mmHg in diabetics patients). All patients who have reached their BP target will be considered as having met the primary endpoint and this visit will be considered as the final visit.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, with essential hypertension, stage I-II, naïve or not controlled with monotherapy.

Exclusion Criteria:

* BP> 180/110 mmHg
* Pregnant or nursing women
* Hypertensive encephalopathy or cerebrovascular accident, transient ischemic - cerebral attack, myocardial infarction, unstable angina, coronary bypass surgery, percutaneous coronary intervention within 6 month
* K <3.5 mEq/L or ≥ 5 mEq/L
* Renal impairment
* Hypersensitivity to HCTZ or Aliskiren or angioedema due to ACE-I or ARB
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The proportion of patients in whom BP control was achieved at the study end point | 16 weeks

SECONDARY OUTCOMES:
The proportion of patients in whom BP control was reached before the addition of HCTZ (ie, at the pre-HCTZ end point | 8 weeks
Percentage of patients achieving overall BP, DBP, an SBP control rate at week 4, 8, 12 and 16. | 16 weeks
Change in msSPA and msDBP from baseline to different time points | 4,8,12 and 16 weeks
Safety of Aliskiren therapy at different time points | 4,8,12 and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Venezuela (7):
  - Investigative Site, Bolíva
  - Investigative Site, Carabobo
  - Investigative Site, Caracas
  - Investigative Site, Edo Zulia
  - Investigative Site, Estado Monagas
  - Investigative Site, Falcón
  - Investigative Site, Maracaibo Estado Zulia